CLINICAL TRIAL: NCT05252117
Title: Blocking the Uterovaginal Plexus With Artacine for Placement of the Intra Uterine Device
Brief Title: Uterovaginal Plexus Block With Articaine for Intrauterine Device Placement Patients Who Are Indicated for the Use of Copper IUD as a Contraceptive Method Will be Invited to Participate in This Research.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Thaise de Melo Nery, Principal investigator, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2022-01-30; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Contraception; IUD; Anesthesia, Local
MeSH Terms: interventions — Carticaine; Mepivacaine

STUDY DESIGN:
Intervention Model Description: Patients will be allocated, according to randomization into one of two groups, after gynecological evaluation at the Gynecology Outpatient Clinic of Hospital das Clínicas Samuel Libânio, in Pouso Alegre. They will be informed about the study and invited to participate and, accepting, signing the Informed Consent Form. Randomization will be followed to define which drug will be used in the patient who will undergo the procedure determined by the study, in a modified lithotomy position, always by the same examiner.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Articaine 4% (Experimental): With the patient in the lithotomy position, asepsis of the thighs, vulva and vagina will be performed with aqueous chlorhexidine; insertion of vaginal speculum; puncture in the uterine cervix, at the 12h point, injecting 1.8 ml of articaine. After a latency of five minutes, the procedure to insert the IUD will start with clamping the cervix at 12 hours with the Pozzi clamp, followed by rectification of the uterus and hysterometry with the hysterometer. After confirming the hysterometry, the IUD will be inserted with its own applicator and the excess wire will be cut.
  Interventions: Drug: Articaine Hydrochloride 40 MG/ML
- Mepivacaíne 3% (Experimental): With the patient in the lithotomy position, asepsis of the thighs, vulva and vagina will be performed with aqueous chlorhexidine; insertion of vaginal speculum; puncture in the uterine cervix, at the 12h point, injecting 1.8 ml of Mepivacaine. After a latency of five minutes, the procedure to insert the IUD will start with clamping the cervix at 12 hours with the Pozzi clamp, followed by rectification of the uterus and hysterometry with the hysterometer. After confirming the hysterometry, the IUD will be inserted with its own applicator and the excess wire will be cut.
  Interventions: Drug: Mepivacaine

INTERVENTIONS:
Drug: Articaine Hydrochloride 40 MG/ML — Analysis of uterovaginal plexus block with articain for intrauterine device placement
  Arms: Articaine 4%
Drug: Mepivacaine — Analysis of uterovaginal plexus block with mepivacaine for intrauterine device placement
  Arms: Mepivacaíne 3%

SUMMARY:
The use of intrauterine device (IUD) in Brazil is still not very significant and one of the reasons is the fear of feeling pain during its insertion procedure. Articaine is an amide-linked local anesthetic, its plasma half-life is shorter than that of most other amide-type anesthetics, which makes it theoretically favorable in relation to systemic toxicity.

DETAILED DESCRIPTION:
Currently, 55% of pregnancies in Brazil are classified as unwanted and approximately only 3% of women use long-term contraception. Intrauterine devices (IUD) are among the most effective long-acting reversible contraceptives, with a failure rate ranging from 0.6 to 0.8% and a duration of 10 years, In Brazil, copper, copper with silver, mirena (levonorgestrel 52mg) and Keelyna (levonorgestrel 13.5mg) IUDs are available. The copper device (T380A) is provided free of charge by the municipal health department. In this sense, they are appropriate methods for most women, including nulliparous women.

Copper IUD, a non-hormonal contraceptive method, causes an inflammatory reaction in the endometrium, with important histological and biochemical changes (increase in cytotoxic cytokines), which interfere with the normal physiology of spermomigration, egg fertilization and blastocyst implantation. Copper ions interfere with vitality and sperm motility, harming them, and also decrease the egg's survival in the genital tract. Copper is responsible for an increase in the production of prostaglandins and inhibition of endometrial enzymes. These changes adversely affect sperm transport so that fertilization rarely occurs. Ovulation is not affected in copper IUD users. Thus, according to available scientific data, copper-containing IUDs act not only in the uterine cavity, but also outside it, interfering with various stages of the reproductive process.

The use of an IUD requires insertion by a duly qualified professional. It is essential that the patient is healthy. Therefore, it is essential: normal gynecological examination; oncotic colpocytology within normal limits; absence of vaginitis, infectious cervicitis, acute or chronic pelvic inflammatory disease, uterine malformations; absence of heart disease, hematological diseases, especially hemorrhagic ones, immune deficiencies; not be pregnant.

The IUD insertion technique is described as follows: Patient in lithotomy position, performing a bimanual vaginal touch and correct assessment of the position of the uterus; vaginal speculum introduction with good exposure of the cervix; antisepsis; clamping of the anterior labrum of the cervix with Pozzi clamp; performing hysterometry - reassessing uterine position and cavity size; place, only at this moment, the IUD inside the applicator shirt; note that the horizontal branches are in the same direction as the lateral diameter of the uterus; insert the applicator with the IUD into the uterus until you feel it has reached the uterine fundus; hold the applicator plunger and pull the shirt, causing the device to extrude into the uterine cavity; carefully remove the applicator; cut the strands, which were left in the vagina, about 2 cm from the external orifice of the cervix. The fear of feeling pain during insertion is one of the reasons for the low acceptance of the method in Brazil. The pain reported by women who undergo IUD insertion without sedation occurs when clamping the cervix, so that the gynecologist can rectify the uterus and when the hysterometer and later the IUD pass through the cervix. Innervation to the uterus and cervix is provided via S2-S4, and visceral pain via afferent fibers from T10-L1. It is believed that the anesthetic instilled in the uterus acts on these nerve endings.

The phenomenon of pain and its concept has often been the subject of several scientific studies. According to the International Association for the Study of Pain, this phenomenon is characterized by an unpleasant sensory and emotional experience, in which there is the perception of a harmful stimulus associated with actual or potential tissue damage.

Anesthesia is the loss of sense or sensation, and local anesthetics are substances that, in contact with a nerve fiber, have the property of interrupting all modalities of nerve inflow. Properly applied local anesthetics are a useful tool to effect a reversible blockade of stimulus conduction (action potential) by nerve fibers (sensory and motor) in the vicinity where they are administered. Local anesthetics are divided into two broad groups: esters and amides. The main structural difference between esters and amides is the bond between the side chain and the saturated ring. When compared to esters, amides are more stable (they can be autoclaved without changing their properties), their hypersensitivity reactions are very rare and, as they undergo hepatic metabolism, they have a longer duration of action.

Articaine, an amide-linked local anesthetic, was approved for use in Brazil in 1999 and has been available in Europe since 1976 and in Canada since 1984. Its plasma half-life is shorter than that of most other amide-type anesthetics. like the other factors, they would be theoretically favorable in relation to systemic toxicity. The potential side effect of the administration of large doses of articaine is methaemoglobinaemia, a reaction perceived after accidental intravenous administration, when performing regional anesthesia. It is a drug biotransformed by plasma and tissue cholinesterases and generates an inactive metabolite, with irrelevant cardiac and neurological toxicity. Because of this, it is an appropriate drug to be used in patients with hepatic and renal dysfunction. Articaine is contraindicated in patients with idiopathic or congenital methaemoglobinaemia, anemia, or cardiac or respiratory failure evidenced by hypoxia.

ELIGIBILITY:
Inclusion Criteria:

- Female patients, aged between 20 and 40 years

Exclusion Criteria:

* Diabetes (type I or II)
* Chronic Kidney
* Urogenital infections
* Psychiatric disesas
* Surgery during the study period

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged 20 to 40 years for insertion of the intrauterine device
Enrollment: 240 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 15 minutes
  analog verbal scale numbered from 0 to 3

SECONDARY OUTCOMES:
sociodemographic data | 10 minutes
  data collection questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade do Vale do Sapucaí, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD under discussion